CLINICAL TRIAL: NCT00697996
Title: A Prospective Open-Labeled Randomized Study of Rituximab Versus Standard of Care, for Treatment of Acute Allograft Rejection in Pediatric Renal Transplantation
Brief Title: Rituximab for Pediatric Renal Transplant Rejection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Genentech and Biogen IDEC (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-06102008-1196
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Rituximab; Graft Rejection

INTERVENTIONS:
Drug: Rituximab for transplant rejection

SUMMARY:
Rituximab will be tested for its safety and potential efficacy in treating B cell dense renal allograft rejection episodes in children receiving renal transplants at Stanford University

DETAILED DESCRIPTION:
Twenty kidney transplant recipients who are being cared for at Stanford University and UCLA and are between the ages of 2-21, can be considered for participation in this research if they are having an acute rejection episode. After a biopsy is done and the diagnosis of acute rejection is made, ten patients will be randomly enrolled in the group to be treated with Rituximab and steroid pulses. Ten children will be enrolled as the control group, receiving standard of care for acute transplant rejection.

Assignment will be based on a 1:1 randomization scheme. That means two patients will be assigned to the group of patients receiving steroid pulsing and 4 doses of Rituximab. The third patient would be assigned to the group receiving steroid pulses and adjustment in immunosuppression medications which is the standard of care at Stanford University.

The dose of Rituximab that will be given is 375 mg/m2 and is administered through an IV. Additional doses of Rituximab will be administered on a weekly basis. A total of four doses will be given.

If the acute rejection does not resolve by one-week, patients in both groups have the option of receiving polyclonal antibody therapy.

ELIGIBILITY:
Inclusion Criteria:Patients must meet the following inclusion criteria to be eligible for study entry:

* Pediatric renal allograft recipients aged 2-21 years with biopsy proven acute rejection episodes.
* Able and willing to give written informed consent and comply with the requirements of the study protocol (patients >18 years of age or parents)
* Greater than 30% decline in baseline renal function as indicated by a rise in the serum creatinine.
* Adequate liver function, as indicated by AST or ALT <2x upper limit of normal unless related to primary disease.
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.

Exclusion Criteria:Patients will be excluded from the study based on the following criteria:

* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of HIV (positive HIV, HIV conducted during screening if applicable)
* History of Hepatitis B and/or Hepatitis C (Hep B/C at screening)
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids (>10mg/day) or unstable steroid dose in the past 4 weeks.
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of psychiatric disorder
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2007-08

PRIMARY OUTCOMES:
Rituximab safety in pediatric patients

SECONDARY OUTCOMES:
resolution fo graft rejection

CONTACTS AND LOCATIONS:
Overall Officials: Minnie M. Sarwal, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States